CLINICAL TRIAL: NCT03187691
Title: An Open Label Phase II Clinical Study to Evaluate the Safety and Pharmacokinetics of Oral Encochleated Amphotericin B (CAMB/MAT2203) for Antifungal Prophylaxis in Patients Undergoing Induction Chemotherapy for Acute Myelogenous (AML) and Lymphoblastic Leukaemia (ALL)
Brief Title: Safety and PK of Oral Encochleated Amphotericin B (CAMB/MAT2203) for Antifungal Prophylaxis in Patients Undergoing Induction Chemotherapy for Acute Myelogenous and Lymphoblastic Leukaemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Protocol redundancy
Sponsor: Matinas BioPharma Nanotechnologies, Inc. (Industry)
Collaborators: University of Cologne (Other); The Clinical Trials Centre Cologne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MB-70006
Record Dates: First submitted 2017-05-31; First posted 2017-06-15 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Non-randomized, open uncontrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CAMB 200 mg (Experimental): 200 mg CAMB (MAT2203) Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)
- CAMB 400 mg (Experimental): 400 mg CAMB (MAT2203) Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)
- CAMB 800mg (Experimental): 800 mg CAMB (MAT2203) Oral Amphotericin B
  Interventions: Drug: Oral Encochleated Amphotericin B (CAMB)

INTERVENTIONS:
Drug: Oral Encochleated Amphotericin B (CAMB) — Lipid-crystal nano-particle formulation amphotericin B
  Other Names: MAT2203

SUMMARY:
A Non-randomized, prospective , multicenter, open uncontrolled study in patients with acute myelogenous (AML) or lymphoblastic leukaemia (ALL)

DETAILED DESCRIPTION:
This is an open label phase II clinical study to evaluate the safety and pharmacokinetics of oral encochleated Amphotericin B (CAMB/MAT2203) for prevention of invasive fungal infections in approximately 30 patients undergoing induction therapy for AML/ALL.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML/ALL receiving chemotherapy inducing neutropenia < 500 cells/mm3
* Able to have all screening tests done to allow for study drug administration no later than 5 days after start of chemotherapy
* Sign informed consent
* ≥ 18 years of age

Exclusion Criteria:

* Known hypersensitivity to amphotericin B, specifically anaphylactic reaction
* Fungal induced fever (≥ 38°C)
* Proven, possible or probably invasive fungal infection in previous 12 months
* Serum galactomannan index (GMI)≥ 0.5 at screening
* Pulmonary infiltrates at screening
* Current treatment with amphotericin B
* Sever comorbidity other than underlying haematological disease
* Prolongation of corrected QT interval
* History of convulsion
* Pregnant or breastfeeding
* Females of childbearing potential who do not practice sexual abstinence or who do not agree to use appropriate contraceptive methods
* Presence of hepatic disease
* Total bilirubin > 3 x upper limit of normal
* Age-adjusted creatinine clearance < 30 mL/minute
* Participating in any other clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 35 days
  Safety assessments include laboratory tests, vital signs, physical exam and ECG

SECONDARY OUTCOMES:
Population pharmacokinetic (PK) analysis | 35 days
  PK parameter for Time to maximum concentration (Tmax)
Population pharmacokinetic (PK) analysis | 35 days
  PK parameter for Peak plasma concentration (Cmax)
Population pharmacokinetic (PK) analysis | 35 days
  PK parameter for Area under the plasma concentration time curve (AUC)
Efficacy analysis for time to clinical symptoms of fungal infection | 35 days
  Clinical symptoms of fungal infections include evaluation of respiratory symptoms, sinuses, skin.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cornely, MD, Principal Investigator — University of Cologne

IPD SHARING:
Plan to Share IPD: No